CLINICAL TRIAL: NCT04677556
Title: Comparison Between Continuous Positive Airway Pressure (CPAP) and Non Invasive Positive Pressure Ventilation (NiPPV) in Bronchiolitis Under Non- Invasive Ventilation
Brief Title: Work of Breathing in Bronchiolitis Under Non-invasive Ventilation
Acronym: BRONCHIO-VNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP200838; 2020-A01419-30 (Other: ID-RCB Number)
Record Dates: First submitted 2020-12-03; First posted 2020-12-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Severe Viral Bronchiolitis
Keywords: Severe acute bronchiolitis; Non-invasive positive pressure ventilation; Continuous positive airway pressure; Work of breathing; Pediatric intensive care
MeSH Terms: conditions — Bronchiolitis, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Severe acute bronchiolitis (Other): Infants under 6 months admitted in Pediatric Intensive Care Unit for a severe acute bronchiolitis needing NIV (modified Woof clinical asthma score (WCAS) >4 and/or hypercapnic acidosis (pH<7,3 and/or pCO2>50mmHg)
  Interventions: Other: Esogastric pressures measurement

INTERVENTIONS:
Other: Esogastric pressures measurement — Catheter placement : at least 2 hours after and within 24 hours following the initial ventilation support establishment (CPAP or NiPPV according to usual practice and clinical conditions). 2 periods of measurements : with the initial and with the 2nd ventilation support using a cross-over for each patient. For each period, the first serie of measurements will be carried out without modifying the settings of the support ( "clinical" setting), and the second one using esogastric pressures by adjusting the settings of the ventilation support in order to obtain an optimal normalization or reduction of the amplitude of the Pes and Pdi deltas ("physiological" setting). 5 minutes of spontaneous breathing with/without oxygen between period 1 and 2 (depending on the patient's conditions). All measurements will be performed for 5 minutes after a 15 minutes quiet breathing. After measurements, the optimal respiratory support will be continued.

SUMMARY:
Severe acute viral bronchiolitis is the leading cause of pediatric intensive care admission. The first-line recommended ventilation support is continuous positive airway pressure (CPAP), which reduces the work of breathing (WOB) and improves gas exchange. Although Non invasive Positive Pressure Ventilation (NiPPV) is increasingly used in case of CPAP failure to avoid intubation, no study has yet evaluated if this support could effectively reduce the effort of breathing.

Our hypothesis is that NiPPV could reduce WOB more effectively than CPAP alone, and might lead to reduce intubation in the most severe bronchiolitis.

The purpose of this study is to compare WOB between CPAP and NiPPV, thanks to esophageal pressure measurement, in infants hospitalized for severe acute bronchiolitis.

DETAILED DESCRIPTION:
Severe acute viral bronchiolitis is the leading cause of pediatric intensive care admission. The first-line recommended ventilation support is non invasive ventilation (NIV) with continuous positive airway pressure (CPAP), which has been proved to reduce the work of breathing (WOB) and improve gas exchange. Non invasive Positive Pressure Ventilation (NiPPV) is increasingly used in case of CPAP failure to avoid intubation. Nevertheless, no study has ever evaluated its effectiveness on the discharge of respiratory muscles in severe bronchiolitis.

Measurement of esophageal and gastric pressures with an esogastric catheter allows an estimation of WOB thanks to the calculation of the esophageal pressure-time product (PTPes), and a calculation of the transdiaphragmatic pressure (Pdi) as the difference between gastric and esophageal pressures. This minimally invasive technique can be used at the bedside to assess the efficacy of ventilation support and is now increasingly used in Intensive Care Units to assist ventilation-targeted strategies.

Our hypothesis is that NiPPV could reduce WOB more effectively than CPAP alone, and might lead to reduce intubation in the most severe bronchiolitis.

The main purpose of this study is to compare PTPes/min between CPAP and NiPPV in infants hospitalized for severe acute bronchiolitis.

Secondary objectives are i) to compare other parameters of WOB, gas exchanges and breathing pattern in both ventilator supports ii) to compare the rate of patient-ventilator asynchronies in 2 different setting of NiPPV ("clinical" and "physiological") iii) to assess if NiPPV is associated with reduced intubation rate, time under sedation and ventilation, and length of hospitalization as compared to CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of bronchiolitis
* Need for non-invasive ventilation support (NiPPV or CPAP) with a modified Wood clinical asthma score (m-WCAS)> 4 and / or hypercapnic acidosis (pH <7.3 and / or pCO2> 50mmHg)
* Written parental informed consent

Exclusion Criteria:

* Contraindication to nasogastric tube (recent surgery of the esophagus, esophageal malformation at risk of perforation, severe coagulopathy)
* Absolute or relative contraindication to NIV

  * Respiratory collapse: coma (GCS <12) and / or more than 3 apneas per hour with bradycardia <90 / min and / or SpO2 <90%
  * Pneumothorax
* Preexisting disorder that may influence WOB

  * Neuromuscular disease
  * Chronic respiratory failure already under NIV or tracheostomy at home
* No social security

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
Esophageal pressure-time product per minute (PTPes/min) | 20 minutes
  Esophageal pressure-time product per minute (PTPes/min) is calculated by the area under the curve of the Pes during inspiration, expressed in cmH2O.s / min.
  The PTPes/min will be measured under CPAP (" clinical" and "physiological" setting) and under NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.

SECONDARY OUTCOMES:
Respiratory rate (RR) | 20 minutes
  Breathing pattern Paramaters will be measured under CPAP ("clinical" and "physiological" setting) and NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.
Heart rate (HR) | 20 minutes
  In pulses per minute Breathing pattern Paramaters will be measured under CPAP ("clinical" and "physiological" setting) and NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.
Inspiratory time (Ti) | 20 minutes
  In sec Breathing pattern Paramaters will be measured under CPAP ("clinical" and "physiological" setting) and NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.
Total respiratory cycle time (Ttot) | 20 minutes
  In sec Breathing pattern Paramaters will be measured under CPAP ("clinical" and "physiological" setting) and NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.
Tidal volume (Vt) | 20 minutes
  In mL Breathing pattern Paramaters will be measured under CPAP ("clinical" and "physiological" setting) and NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.
Gas exchange | 3 hours
  SpO2 and PtcCO2, in mmHg will be continuously monitored thanks to a pulse oxymeter and transcutaneous capnography (SenTecTM) for 3 hours
Modified Wood's Clinical Asthma Score (m-WCAS) | At inclusion and at the end of the measurements, i.e. 3 hours from inclusion
  Modified Wood's Clinical Asthma Score (m-WCAS) is a respiratory failure score that includes 3 levels of gravity corresponding to 5 respiratory distress clinical signs. Values ranged from 0 (best score) to 10 (worst score)
PEdiatric Logistic Organ Dysfunction-2 score (PELOD-2) | At inclusion and at the end of the measurements, i.e. 3 hours from inclusion
  Pediatric logistic organ dysfunction score is a specific pediatric multiple organ dysfunction score that includes 10 variables corresponding to 5 organ dysfunctions. Values extend from 0 (best outcome) to 33 (worst outcome).
Work of breathing | 20 minutes
  Esophageal pressure delta (ΔPES, normal between 5 and 8 cmH2O) Transdiaphragmatic pressure delta (ΔPdi). The Pdi is obtained by subtracting the Pes from the Pgas Pressure-time product of the diaphragm per minute (PTPDdi/min).
  Paramaters will be measured under CPAP (" clinical" and "physiological" setting) and under NiPPV (" clinical" and "physiological" setting) during a period of quiet breathing of 5 minutes.
Need for intubation | Through study completion, an average of 2 years
Number of days under sedation by Midazolam IV or per os upon hospital discharge | Through study completion, an average of 2 years
Number of days under NIV | Through study completion, an average of 2 years
Number of days under invasive ventilation | Through study completion, an average of 2 years
Number of days in intensive care unit | Through study completion, an average of 2 years
Number of days in hospitalization | Through study completion, an average of 2 years
Patient-ventilator asynchronies (under NiPPV) | Through study completion, an average of 2 years
  Patient-ventilator asyncrhonies will be analyzed using the flow and pressure curves of the ventilator and the patient (Pes), then classified into 4 groups:
  * auto-triggering (cycle delivered by the ventilator without patient's inspiratory effort),
  * double triggering (2 successive cycles delivered by the ventilator for a single inspiratory effort of the patient),
  * wasted effort (patient inspiratory effort not followed by a cycle delivered by the ventilator),
  * daly asynchronies (advance or delay of the cycle delivered by the ventilator compared to the start of the patient's inspiration or expiration) The percentage of patient-ventilator asynchronies will be analyzed under NiPPV ("clinical" setting and "physiological" setting) during a period of quiet breathing of 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Meryl VEDRENNE-CLOQUET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Brigitte FAUROUX, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vedrenne-Cloquet M, Khirani S, Griffon L, Collignon C, Renolleau S, Fauroux B. Respiratory effort during noninvasive positive pressure ventilation and continuous positive airway pressure in severe acute viral bronchiolitis. Pediatr Pulmonol. 2023 Jul;58(7):2000-2008. doi: 10.1002/ppul.26424. Epub 2023 Apr 25. PMID 37097049